CLINICAL TRIAL: NCT04788849
Title: Extended VALidation of HUman Papillomavirus Assays and Collection DEvices for HPV Testing on Self-samples and First-void Urine Samples
Brief Title: Extended VALidation of HUman Papillomavirus Assays and Collection DEvices for HPV Testing on Self-samples
Acronym: Ext-VALHUDES
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Collaborators: Becton, Dickinson and Company (Industry); COPAN ITALIA SPA (Unknown); Sciensano (Other Government); Istituto Europeo di Oncologia (Other); Università degli Studi di Sassari (Other); ATS Sardegna (Unknown)
Responsible Party: Sponsor
Other Study IDs: UMilanoBicocca&BD/Copan
Record Dates: First submitted 2021-03-03; First posted 2021-03-09 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2023-05

CONDITIONS: Cervical Intraepithelial Neoplasia Grade 2/3; Carcinoma Cervix
Keywords: Self-Sampling; HPV testing; Diagnostic Test Accuarcy; Cervical Cancer Screening; Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Vaginal, urine and cervical samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Women referred to colposcopy: Three sample types (urine, vaginal and cervical) will be collected from all enrolled women.
  Interventions: Diagnostic Test: BD Onclarity™ HPV assay

INTERVENTIONS:
Diagnostic Test: BD Onclarity™ HPV assay — Women will be asked to self-collect first-void urine using Copan's UriSponge™ 8E031S100 and vaginal swabs using Copan's FLOQSwabs® 5E089N. All samples will be tested with BD Onclarity™ HPV assay. HPV test results on self-collected samples will be compared to those obtained when testing clinician-collected cervical sample
  Other Names: Copan's FLOQSwabs® 5E089N; Copan's UriSponge™ 8E031S100

SUMMARY:
The "Extended VALHUDES" study is a Clinical Performance / Diagnostic Test Accuracy Study that aims to extend validation, achieved as part of the "Belgian VALHUDES", of HPV testing using BD Onclarity on samples collected using Copan's devices for dry self-sampling of vaginal material and for first-void urine: FLOQSwab® 5E089N and UriSponge™.

DETAILED DESCRIPTION:
Women accessing the Colposcopy Centres for a colposcopy examination and fulfilling the selection criteria will be asked, after written informed consent, to self-collect a first-void urine (with UriSponge™ 8E031S100 device) and a vaginal sample (with FLOQSwab® 5E089N device), prior to undergoing colposcopy. Just before colposcopic examination, a clinician will also collect a cervical sample using a Cervex-Brush.

A colposcopy-targeted biopsy or histology following excisional treatment of a cervical precancer lesion will be undertaken if appropriate. The colposcopy and/or histological findings will be used as the gold standard. In case of normal satisfactory colposcopic findings without biopsy taking, colposcopy will provide the study outcome.

Virological accuracy of HPV testing using: [a] BD Onclarity on FLOQSwab® 5E089N vaginal self-samples, [b] BD Onclarity on UriSponge™ 8E031S100 urine specimens, will be compared to BD Onclarity testing on a cervical samples collected by a clinician.

ELIGIBILITY:
Inclusion Criteria:

* Women, referred to colposcopy due to abnormal Pap-test result, who agree to participate in the study by signing an informed consent form

Exclusion Criteria:

* Women younger than 25 or older than 64 years of age
* Hysterectomized women
* Women with known pregnancy
* Non-consenting women
* Women that are not able to understand and/or sign the informed consent.

Ages: 25 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with a recent history of abnormal Pap smear who are referred to colposcopy in one of the 2 Italian Colposcopy Centres:
  * Istituto Europeo di Oncolgia (IEO), Milan
  * Coordinamento Consultori Familiari, ATS Sardegna
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Analytical performance and Clinical accuracy | One day, with possible extension if excision biopsy is planned based on the coloposcopy/histology outcome of tissue specimens collected at the enrolment visit.
  Concordance of the presence of HPV and of the partial and extended HPV genotyping results applied on self- and clinician-collected samples.

SECONDARY OUTCOMES:
Women's Acceptance and Preferences regarding urine collection, vaginal self-sampling or cervical sample collection by a clinician. | One day
  Acceptance and preferences regarding urine collection, vaginal self-sampling or clinicians' collected cervical samples will be assessed through a questionnaire administered to participating women at the time of colposcopy. The questionnaire will allow to determine the percentage of women expressing a preference for urine collection and/or vaginal self-sampling over clinicians' collected cervical samples.

CONTACTS AND LOCATIONS:
Overall Officials: Clementina E. Cocuzza, MD, PhD, Principal Investigator — School of Medicine and Surgery, University of Milano-Bicocca
Locations (2):
- Italy (2):
  - IEO European Institute of Oncology, Milan
  - Coordinamento Consultori Familiari ASSL Sassari, Sassari

IPD SHARING:
Plan to Share IPD: No
Study protocol and results have been published:
  Martinelli M, Latsuzbaia A, Bonde J, Pedersen H, Iacobone AD, Bottari F, Piana AF, Pietri R, Cocuzza CE, Arbyn M; Extended Valhudes Study Group. Performance of BD Onclarity HPV assay on FLOQSwabs vaginal self-samples. Microbiol Spectr. 2024 Mar 5;12(3):e0287223. doi: 10.1128/spectrum.02872-23. Epub 2024 Feb 7. PMID: 38323823; PMCID: PMC10913526.

REFERENCES:
- [Background] Arbyn M, Peeters E, Benoy I, Vanden Broeck D, Bogers J, De Sutter P, Donders G, Tjalma W, Weyers S, Cuschieri K, Poljak M, Bonde J, Cocuzza C, Zhao FH, Van Keer S, Vorsters A. VALHUDES: A protocol for validation of human papillomavirus assays and collection devices for HPV testing on self-samples and urine samples. J Clin Virol. 2018 Oct;107:52-56. doi: 10.1016/j.jcv.2018.08.006. Epub 2018 Aug 22. PMID 30195193
- [Background] Arbyn M, Verdoodt F, Snijders PJ, Verhoef VM, Suonio E, Dillner L, Minozzi S, Bellisario C, Banzi R, Zhao FH, Hillemanns P, Anttila A. Accuracy of human papillomavirus testing on self-collected versus clinician-collected samples: a meta-analysis. Lancet Oncol. 2014 Feb;15(2):172-83. doi: 10.1016/S1470-2045(13)70570-9. Epub 2014 Jan 14. PMID 24433684
- [Background] Arbyn M, Smith SB, Temin S, Sultana F, Castle P; Collaboration on Self-Sampling and HPV Testing. Detecting cervical precancer and reaching underscreened women by using HPV testing on self samples: updated meta-analyses. BMJ. 2018 Dec 5;363:k4823. doi: 10.1136/bmj.k4823. PMID 30518635